CLINICAL TRIAL: NCT06915935
Title: Study on the Epidemiological Characteristics of Osteoporosis and the Diagnostic Significance of Bone Metabolic Biochemical Markers in the Elderly Population of Shandong Province
Brief Title: Epidemiological Study of Osteoporosis in the Elderly Population of Shandong Province
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL2024022
Record Dates: First submitted 2025-03-28; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis; Osteoporosis (Senile)
Keywords: osteoporosis; epidemiology; elderly; Biochemical indexes of bone metabolism
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- osteoporosis: Based on the economic development level, population composition, geographical location, cost-effectiveness and feasibility of the program, a cross-sectional survey was conducted to investigate the community population in Shandong Province from August 1, 2023 to January 31, 2026, covering cities and rural areas in the east, west, south, north and middle prefecture-level cities in 10 regions. The inclusion population was residents ≥65 years of age who had lived in the area for more than 6 months in the past 1 year, and the exclusion criteria were cognitive impairment or mental illness.
  Interventions: Radiation: dualenergy X-ray absorptiometry

INTERVENTIONS:
Radiation: dualenergy X-ray absorptiometry — Dual-energy X-ray Absorptiometry (DXA) is an accurate, safe, and rapid bone mineral density measurement method that is widely used in the diagnosis of osteoporosis and the assessment of fracture risk. The principle is based on the difference in absorption of different energy X-rays in bone and soft tissue, and bone mineral content (BMC) and bone mineral density (BMD) are obtained through mathematical calculations. DXA is commonly used to measure bone mineral density in the lumbar spine, femoral neck, and forearm, and to assess the degree of osteoporosis using a T score, where T ≤ -2.5 is defined as osteoporosis. Due to the advantages of high precision, low radiation dose and convenient operation, DXA is considered as the gold standard for clinical bone mineral density detection.

SUMMARY:
At present, there is little epidemiological information on osteoporosis in the elderly population of Shandong Province, especially the lack of systematic research on the role of bone metabolism and biochemical indicators in the diagnosis and prognosis of osteoporosis in the elderly population of Shandong Province. The group intends to conduct a study on the epidemiological characteristics of osteoporosis patients and the significance of bone metabolism biochemical indexes in the diagnosis and prognosis of osteoporosis in elderly people in Shandong Province, which includes 1) assessing the prevalence of osteoporosis and the risk factors associated with osteoporosis in the community population, and 2) exploring the role of bone metabolism biochemical indexes in the diagnosis and prognosis of osteoporosis in the hospitalised population. Expected outcomes include the establishment of a database of community and inpatient populations in Shandong Province, publication of research papers, and participation in academic conferences at home and abroad. The database will collect and organise data on osteoporosis in the community and inpatient osteoporosis in Shandong Province, and provide support for subsequent data analysis and research.

ELIGIBILITY:
Inclusion Criteria:

* Residents ≥65 years of age who had lived in the area for more than 6 months in the past 1 year

Exclusion Criteria:

* People with cognitive impairment or mental illness

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: According to the level of economic development, population composition, geographical location, cost-effectiveness and feasibility of the program, a total of 10 regions covering five prefecture-level cities in east, west, south, north and middle of Shandong Province were selected to investigate the community population in Shandong Province from August 1, 2023 to January 31, 2026. The inclusion population was residents ≥65 years of age who had lived in the area for more than 6 months in the past 1 year, and the exclusion criteria were cognitive impairment or mental illness.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | baseline
  Bone Mineral Density (BMD) refers to the mineral content per unit area or unit volume of bone tissue, usually expressed in g/cm², and is an important indicator to measure bone strength and assess the risk of osteoporosis.

SECONDARY OUTCOMES:
Numerical Rating Scale | baseline
  The patient's pain intensity is evaluated by Numerical Rating Scale. Patients are required to select a number to represent the pain intensity according to their own feelings within the numerical range of 0 to 10, in which 0 represents no pain and 10 represents extremely severe pain.
Grip strength test | baseline
  Grip strength examination is a common method to evaluate hand muscle strength and overall muscle strength, which is widely used in rehabilitation assessment, nutritional status judgment and health monitoring of the elderly.

CONTACTS AND LOCATIONS:
Locations (1):
- Community/rural health service centres, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided